CLINICAL TRIAL: NCT05600595
Title: The Evaluation of Eustachian Tube Function and Its Influencing Factors After Snoring in Children
Brief Title: The Evaluation of Eustachian Tube Function and Its Influencing Factors After Snoring Operation in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Xiaolan People's Hospital of Zhongshan City (Unknown)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-350-01
Record Dates: First submitted 2022-10-27; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Adenoidectomy; Tonsillectomy; Eustachian Tube Dysfunction
Keywords: Eustachian Tube Dysfunction; Snoring in children
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Operation for snoring in children — Tonsillectomy and/or adenoidectomy

SUMMARY:
This study aims to evaluate and screen out the factors related to the improvement of eustachian tube function after adenoidectomy and/or tonsillectomy, so as to guide the treatment of children's eustachian tube function before and after operation, and provide the treatment direction and methods for diseases related to eustachian tube dysfunction for people with adenoid hypertrophy and/or tonsil hypertrophy complicated with ETD.

DETAILED DESCRIPTION:
This study aims to analyze the changes of eustachian tube function in children with snoring and eustachian tube dysfunction before and after snoring surgery, and to evaluate and screen out the related factors related to the improvement of eustachian tube function after snoring surgery. The patients who were admitted to hospital and diagnosed as children's snoring complicated with diseases related to eustachian tube dysfunction and planned to undergo surgical treatment for children's snoring should be included, and relevant examinations should be improved, including preoperative nasopharyngoscope, otoscope, acoustic immittance and pure tone audiometry. After snoring operation, he returned to the hospital at 6, 12 and 24 weeks after operation for reexamination of nasopharyngoscope, otoscope, acoustic immittance, pure tone audiometry and TMM. The patients were assessed with ETDQ-7 score, ETS-7 score and VAS score by self-administered questionnaire. The effective risk-related factors were screened out by single factor and multi-factor Logistics regression analysis. To guide the treatment of children's eustachian tube function before and after operation, and to provide the treatment direction and methods for children's snoring diseases complicated with ETD.

ELIGIBILITY:
Inclusion Criteria:

① Age 3-14 years old.

② Patients diagnosed as snoring or adenoid hypertrophy in children, tonsil hypertrophy and chronic tonsillitis who are to be treated by adenoidectomy or tonsillectomy or tonsillectomy;

③ Conform to 1. Symptoms: snoring during sleep, breathing with mouth open, some with apnea, restless sleep, and a few children with hearing loss. 2. Fiberoptic nasopharyngoscopy showed adenoids and/or tonsil hypertrophy. 3. No family history of deafness, no history of ototoxic drugs. 4. No external ear and maxillofacial deformity. 5. The tympanic pressure curve is "C" or "B". 6. No suppurative medium.

Auricular inflammation and tympanic membrane perforation; Adhesive otitis media, cholesteatoma of middle ear.

④ Patients' families cooperated well.

⑤ The patient's guardian volunteered to participate in this study and signed the informed consent form.

Exclusion Criteria:

* Middle ear catheterization or puncture was performed at the same time;

  * Eustachian atresia or cleft lip and palate; There are craniofacial abnormalities or neuromuscular diseases;

    * Benign and malignant tumors of nose or nasopharynx;

      * Other middle ear diseases (suppurative otitis media, tympanic membrane perforation; Adhesive otitis media, middle ear cholesteatoma, etc.); ⑤ Those who can't cooperate; ⑥ Previous tonsil and adenoid surgery; ⑦ Upper respiratory tract infection in recent two weeks; ⑧ Any other circumstances that researchers think should be excluded from this study;

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with snoring complicated with eustachian tube dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Tympanogram | 6 weeks after operation
  Acoustic immittance test

SECONDARY OUTCOMES:
EDTQ-7 symptom score | 6 weeks after operation
  1. Pressure in the ears?
  2. Pain in the ears?
  3. A feeling that your ears are clogged or 'under water'?
  4. Ear symptoms when you have a cold or sinusitis?
  5. Crackling or popping sounds in the ears?
  6. Ringing in the ears?
  7. A feeling that your hearing is muffled
Eustachian tube inflammation | 6 weeks after operation
  Divided into 0=normal, 1=mild, 2=moderate, 3=severe

CONTACTS AND LOCATIONS:
Overall Officials: Hao Xiong, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ockermann T, Reineke U, Upile T, Ebmeyer J, Sudhoff HH. Balloon dilatation eustachian tuboplasty: a clinical study. Laryngoscope. 2010 Jul;120(7):1411-6. doi: 10.1002/lary.20950. PMID 20564474
- [Result] Bluestone CD,Bluestone MB. Eustachian tube：structure，function，role in otitis media. NY：BC Decker，2005
- [Result] Mansour S，Magnan J，Haidar H，et al. Tympanic membrane retraction pocket. Springer International Publishing，2015：17
- [Result] Meyer TA, O'Malley EM, Schlosser RJ, Soler ZM, Cai J, Hoy MJ, Slater PW, Cutler JL, Simpson RJ, Clark MJ, Rizk HG, McRackan TR, D'Esposito CF, Nguyen SA. A Randomized Controlled Trial of Balloon Dilation as a Treatment for Persistent Eustachian Tube Dysfunction With 1-Year Follow-Up. Otol Neurotol. 2018 Aug;39(7):894-902. doi: 10.1097/MAO.0000000000001853. PMID 29912819
- [Result] Alper CM, Luntz M, Takahashi H, Ghadiali SN, Swarts JD, Teixeira MS, Csakanyi Z, Yehudai N, Kania R, Poe DS. Panel 2: Anatomy (Eustachian Tube, Middle Ear, and Mastoid-Anatomy, Physiology, Pathophysiology, and Pathogenesis). Otolaryngol Head Neck Surg. 2017 Apr;156(4_suppl):S22-S40. doi: 10.1177/0194599816647959. PMID 28372527
- [Result] D'Alatri L, Picciotti PM, Marchese MR, Fiorita A. Alternative treatment for otitis media with effusion: eustachian tube rehabilitation. Acta Otorhinolaryngol Ital. 2012 Feb;32(1):26-30. PMID 22500063
- [Result] Schroder S, Lehmann M, Sauzet O, Ebmeyer J, Sudhoff H. A novel diagnostic tool for chronic obstructive eustachian tube dysfunction-the eustachian tube score. Laryngoscope. 2015 Mar;125(3):703-8. doi: 10.1002/lary.24922. Epub 2014 Sep 12. PMID 25215457
- [Result] Cayir S, Hizli O, Kayabasi S, Yildirim G. Eustachian tube dysfunction in sleep apnea patients and improvements afforded by continuous positive airway pressure therapy. Braz J Otorhinolaryngol. 2021 May-Jun;87(3):333-337. doi: 10.1016/j.bjorl.2020.02.003. Epub 2020 Mar 12. PMID 32247766
- [Result] Robison JG, Wilson C, Otteson TD, Chakravorty SS, Mehta DK. Increased eustachian tube dysfunction in infants with obstructive sleep apnea. Laryngoscope. 2012 May;122(5):1170-7. doi: 10.1002/lary.22473. Epub 2012 Feb 16. PMID 22344711
- [Result] Ahmed ST, Lin J, Moskowitz HS, Stupak HD. Can the negative pressures found in obstructive sleep apnea and Eustachian tube dysfunction be related? Am J Otolaryngol. 2021 Jul-Aug;42(4):102993. doi: 10.1016/j.amjoto.2021.102993. Epub 2021 Feb 18. PMID 33640801